CLINICAL TRIAL: NCT00507078
Title: Biomarkers in Obstructive Sleep Apnea Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Eric Kezirian, Associate Professor, Director of Sleep Surgery, University of California, San Francisco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 522315-38198
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Leptin; Homocysteine; C-reactive Protein
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Surgical treatment for OSA

SUMMARY:
Recent years have witnessed major advances in the understanding of the hormonal, metabolic, and biochemical changes that occur in obstructive sleep apnea (OSA). This project evaluates the biomarkers that measure the most significant health impacts of this disorder and creates a specimen bank that will facilitate evaluations of additional biomarkers in the future.

DETAILED DESCRIPTION:
This is a case-control study to examine the relationship between obstructive sleep apnea (OSA) and elevated levels of leptin, homocysteine, and C-reactive protein (CRP) in moderate or severe OSA and control patients. This is followed by a prospective cohort study to examine the relationship between surgical treatment of moderate or severe OSA and serum levels of these biomarkers.

The short-term goals of this study consider the abnormalities in biomarker levels associated with OSA and specific aspects of the disorder as well as whether the changes seen after surgical treatment of OSA mirror those demonstrated after efficacious non-surgical treatment. The long term goals are in two areas: 1) the development of measures to determine which patients require treatment for sleep-disordered breathing and to monitor the effectiveness of therapy, and 2) a deeper understanding of the connection between OSA and its adverse health consequences.

ELIGIBILITY:
Inclusion Criteria:

* OSA group is adults with moderate or severe OSA (apnea >= 15 based on preoperative sleep study) undergoing surgical treatment. Assessment is done prior to surgery.
* Control group is overweight (body mass >25) adults without OSA (apnea-hypopnea index <5 based on sleep study) or other sleep disorders. Assessment is prior to treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Leptin, homocysteine, and C-reactive protein levels. | Before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kezirian, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States